CLINICAL TRIAL: NCT02019667
Title: Phase 2 Clinical Trial of SGS-742 Therapy in Succinic Semialdehyde Dehydrogenase Deficiency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 140033; 14-N-0033 (Other: NIH)
Record Dates: First submitted 2013-12-20; First posted 2013-12-24 (Estimated); Results first posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2018-10

CONDITIONS: Metabolic Disease; Seizures
Keywords: GABA; Seizures; Neurotransmitters
MeSH Terms: conditions — Metabolic Diseases; Seizures | interventions — (3-aminopropyl)(n-butyl)phosphinic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Experimental): Participants with SSADH Deficiency when on placebo for six months
  Interventions: Drug: Placebo
- Study Drug (Experimental): Participants with SSADH Deficiency receiving SGS-742 when on study drug for six months
  Interventions: Drug: SGS-742

INTERVENTIONS:
Drug: SGS-742
  Arms: Study Drug
Drug: Placebo
  Arms: Placebo

SUMMARY:
Objective:

To perform a clinical trial assessing the safety, tolerability and efficacy of the GABA(B) receptor antagonist SGS-742 in patients with SSADH deficiency.

Study Population:

Twenty-two children and adults with SSADH deficiency.

Design:

Double-blind, cross-over, phase II clinical trial.

Outcome Measures:

The primary outcome measures for drug efficacy will be performance on neuropsychological testing and responses to parent questionnaire. The secondary outcome measure will be TMS parameters of cortical excitation and inhibition. The outcome measures for safety will include clinical examination and neuropsychological tests.

DETAILED DESCRIPTION:
Objective:

To perform a clinical trial assessing the safety, tolerability and efficacy of the GABA(B) receptor antagonist SGS-742 in patients with SSADH deficiency.

Study Population:

Twenty-two children and adults with SSADH deficiency.

Design:

Double-blind, cross-over, phase II clinical trial. SGS-742 is a GABA (B) receptor antagonist that has shown to be safe and well-tolerated in clinical trials in adults with cognitive impairment. In addition, preliminary data in the SSADH knockout mouse model suggest efficacy in this specific syndrome. The primary outcome measure will be a change in the Auditory Comprehension subtest of the Neuropsychological Assessment Battery Language Module score; the secondary outcome measure will be a change in cortical excitation and inhibition measured by transcranial magnetic stimulation (TMS). Additional evaluations will include neurological and neuropsychological examinations, magnetic resonance spectroscopy and CSF collection to measure GABA levels. The trial will have a baseline phase in which each patient will undergo a neurological examination and a neuropsychological evaluation. During the subsequent treatment phase, patients will be randomized to SGS-742, supplied by IRIX Pharmaceuticals, and based on weight given a maximum tolerated dose not to exceed 600 mg t.i.d. orally, or placebo, each for 6 months. Patients will then have repeat TMS, neurological and neuropsychological evaluations, followed by cross-over to the alternate treatment arm, and re-evaluation after 6 months.

Outcome Measures:

The primary outcome measures for drug efficacy will be performance on neuropsychological testing and responses to parent questionnaire. The secondary outcome measure will be TMS parameters of cortical excitation and inhibition. The outcome measures for safety will include clinical examination and neuropsychological tests.

ELIGIBILITY:
* INCLUSION CRITERIA
* Aged 4 years or older
* 4-hydroxybutyric aciduria (gamma-hydroxybutyric aciduria) on two separate tests
* Documented succinic semialdehyde dehydrogenase enzyme deficiency
* Patients must have clinical features consistent with SSADH deficiency including developmental delay especially deficit in expressive language, hypotonia, ataxia, seizures, and other neuropsychiatric symptoms including sleep disturbances , attention deficit, anxiety, obsessivecompulsive disorder, and autistic traits
* During the study, women of child-bearing potential must use a reliable method of birth control until one month after the final drug taper is complete.

EXCLUSION CRITERIA

* Current alcohol use (>14 drinks/wk in men and >7 drinks/wk in women or or recreational drug use
* Contraindications to MRI: metal in the body including pacemakers, medication pumps, aneurysm clips, metallic prostheses (including metal pins and rods, heart valves or cochlear implants), shrapnel fragments, permanent eye liner or small metal fragments in the eye that welders and other metal workers may have
* Claustrophobia
* Cannot lie comfortably flat on the back for up to 2h in the MRI scanner
* Patients with a history of other major medical disorders with clinical fluctuations, or requiring therapy that might affect study participation or drug response such as severe depression or psychoses, renal or hepatic disease.
* Patients requiring treatment with drugs known to affect the GABAergic system, including vigabatrin and benzodiazepines.
* Pregnant and lactating women

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-03-31 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara K Inati, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Washington State University, Pullman, Washington

REFERENCES:
- [Background] Al-Essa MA, Bakheet SM, Patay ZJ, Powe JE, Ozand PT. Clinical, fluorine-18 labeled 2-fluoro-2-deoxyglucose positron emission tomography (FDG PET), MRI of the brain and biochemical observations in a patient with 4-hydroxybutyric aciduria; a progressive neurometabolic disease. Brain Dev. 2000 Mar;22(2):127-31. doi: 10.1016/s0387-7604(99)00121-7. PMID 10722966
- [Background] Arnold S, Berthele A, Drzezga A, Tolle TR, Weis S, Werhahn KJ, Henkel A, Yousry TA, Winkler PA, Bartenstein P, Noachtar S. Reduction of benzodiazepine receptor binding is related to the seizure onset zone in extratemporal focal cortical dysplasia. Epilepsia. 2000 Jul;41(7):818-24. doi: 10.1111/j.1528-1157.2000.tb00248.x. PMID 10897152
- [Background] Arnulf I, Konofal E, Gibson KM, Rabier D, Beauvais P, Derenne JP, Philippe A. Effect of genetically caused excess of brain gamma-hydroxybutyric acid and GABA on sleep. Sleep. 2005 Apr;28(4):418-24. doi: 10.1093/sleep/28.4.418. PMID 16171286
- [Derived] Schreiber JM, Wiggs E, Cuento R, Norato G, Dustin IH, Rolinski R, Austermuehle A, Zhou X, Inati SK, Gibson KM, Pearl PL, Theodore WH. A Randomized Controlled Trial of SGS-742, a gamma-aminobutyric acid B (GABA-B) Receptor Antagonist, for Succinic Semialdehyde Dehydrogenase Deficiency. J Child Neurol. 2021 Nov;36(13-14):1189-1199. doi: 10.1177/08830738211012804. Epub 2021 May 20. PMID 34015244
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-N-0033.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited and enrolled in the protocol between March 2014 and October 2017, with assistance from referring physicians in the community and the SSADH foundation. A total of 19 participants were enrolled; 16 completed dosing in both placebo and active drug arms.
Pre-assignment Details: Following a baseline visit, participants were randomized to receive either placebo or study drug for 6 months (Phase 1) followed by 6 months of the alternate treatment (Phase 2). Participants completed a 9-week washout period following each phase of the study.
Groups:
- Placebo First, Then SGS-742: Participants were administered Placebo, followed by a washout period, and then administered SGS-742
- SGS-742 First, Then Placebo: Participants were administered SGS-742, followed by a washout period, and then administered Placebo
Period: First Intervention (6 Months)
Arm/Group | Placebo First, Then SGS-742 | SGS-742 First, Then Placebo
Started | 10 | 9
Completed | 10 | 8
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Washout Period (9 Weeks)
Arm/Group | Placebo First, Then SGS-742 | SGS-742 First, Then Placebo
Started | 10 | 8
Completed | 10 | 8
Not Completed | 0 | 0
Period: 2nd Intervention (6 Months)
Arm/Group | Placebo First, Then SGS-742 | SGS-742 First, Then Placebo
Started | 10 | 8
Completed | 10 | 6
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Physician Decision | 0 | 1
Period: Washout Period (9 Weeks)
Arm/Group | Placebo First, Then SGS-742 | SGS-742 First, Then Placebo
Started | 10 | 6
Completed | 10 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants with SSADH Deficiency who were randomized to receive either SGS-742 or Placebo
Arm/Group | All Study Participants
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 14 (7.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline on the Adaptive Behavior Assessment System (ABAS) Test at the End of the Study Drug and Placebo Treatment Periods
Description: The ABAS questionnaire was completed by the participant's parent or caregiver at the end of each six month treatment period.The ABAS provides a comprehensive picture of adaptive skills across the lifespan. The questionnaire addresses Conceptual, Social and Practical skills including communication, self-direction, use of leisure time, health, safety and self-care. The General Adaptive Composite score ranges from <40 to >160 with a lower score representing lower adaptive behavior. The difference between Placebo and Baseline and Study Drug and Baseline were obtained. These values were averaged across individuals to report a mean and a standard deviation of the baseline-to-treatment period change. The means for each treatment can be compared to have a baseline-adjusted treatment effect interpretation. A positive change represents an improvement in adaptive skills compared with baseline and a negative change represents a decline in adaptive skills compared with baseline.
Time Frame: baseline and six months
Population: The ABAS was not able to be completed for all participants.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Placebo: Participants with SSADH Deficiency when on placebo for six months
  Placebo
- Study Drug: Participants with SSADH Deficiency receiving SGS-742 when on study drug for six months
  SGS-742
Arm/Group | Placebo | Study Drug
Number analyzed (Participants) | 13 | 13
scores on a scale | 5.2 (7.1) | 4.5 (7.5)

2. Secondary Outcome: Change From Baseline of TMS Measurement of Motor Threshold at the End of the Study Drug and Placebo Treatment Periods
Description: Transcranial Magnetic Stimulation (TMS) is a non-invasive technique which applies magnetic pulses to the brain via a coil inducing an electrical current in the brain. Stimulation is typically applied at a sufficient intensity to trigger action potentials in nearby neurons. The motor threshold is defined as the minimum percentage of the stimulator output that evoked a motor evoked potential of more than 50µV in at least 5 out of 10 trials. Motor threshold was measured at the end of the study drug period and the end of the Placebo period. The differences between Placebo and Baseline, and SGS and Baseline were obtained. A decrease from baseline value indicates increased cortical excitability and an increase from baseline value indicates reduced cortical excitability. These values were averaged across individuals to report a mean and standard deviation of this baseline-to-treatment period change. The mean for each treatment can be compared to have a baseline-adjusted treatment effect.
Time Frame: Baseline and Six months
Population: We were unable to obtain Motor Thresholds for all participants at all three timepoints, resulting in different N for each time period. All available data is reported.
Measure: Mean (Standard Deviation); unit: percentage of stimulator output
Arm/Group | Placebo | Study Drug
Number analyzed (Participants) | 16 | 17
percentage of stimulator output | -2 (7.1) | -0.5 (6.8)

3. Secondary Outcome: Change From Baseline of TMS Measurement of Intracortical Facilitation at the End of the Study Drug and Placebo Treatment Periods
Description: Transcranial Magnetic Stimulation (TMS) is a non-invasive technique which applies magnetic pulses to the brain via a coil inducing an electrical current in the brain. Stimulation is typically applied at a sufficient intensity to trigger action potentials in nearby neurons. Intracortical facilitation (ICF) and inhibition (ICI) were studied using a paired stimulus paradigm. The motor threshold (MT) was first established. The conditioning stimulus (70% MT) followed by the test stimulus (120% MT) was delivered at an interstimulus interval (ISI) of 10 ms for ICF. Each run consisted of 10 trials, and the amplitude ratio of the mean conditioned Motor Evoked Potential (MEP) to control MEP was determined. A larger amplitude ratio indicates greater cortical excitability. The differences between Placebo and Baseline, and SGS and Baseline were obtained. These values were averaged across individuals to report a mean.
Time Frame: Baseline and Six months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio of MEP amplitude
Arm/Group | Placebo | Study Drug
Number analyzed (Participants) | 16 | 17
ratio of MEP amplitude | 49.9 (61.9) | 40.5 (50.2)

4. Secondary Outcome: Change From Baseline of TMS Measurement of Short Interval Intracortical Inhibition (Short ICI) at the End of the Study Drug and Placebo Treatment Periods
Description: Transcranial Magnetic Stimulation (TMS) is a non-invasive technique which applies magnetic pulses to the brain via a coil inducing an electrical current in the brain. Stimulation is typically applied at a sufficient intensity to trigger action potentials in nearby neurons. Intracortical facilitation and inhibition were studied using a paired stimulus paradigm. The motor threshold (MT) was first established. The conditioning stimulus (70% MT) followed by the test stimulus (120% MT) was delivered at an interstimulus interval (ISI) of 2 ms for short ICI. Each run consisted of 10 trials, and the amplitude ratio of the mean conditioned Motor Evoked Potential (MEP) to control MEP was determined. A larger amplitude ratio indicates greater cortical excitability. The differences between Placebo and Baseline, and SGS and Baseline were obtained. These values were averaged across individuals to report a mean.
Time Frame: Baseline and Six months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio of MEP amplitude
Arm/Group | Placebo | Study Drug
Number analyzed (Participants) | 16 | 17
ratio of MEP amplitude | 35.5 (123.4) | -11.0 (54.8)

5. Secondary Outcome: Change From Baseline of TMS Measurement of Long Interval Intracortical Inhibition (Long ICI) at the End of the Study Drug and Placebo Treatment Periods
Description: Transcranial Magnetic Stimulation (TMS) is a non-invasive technique which applies magnetic pulses to the brain via a coil inducing an electrical current in the brain. Stimulation is typically applied at a sufficient intensity to trigger action potentials in nearby neurons.Intracortical facilitation and inhibition were studied using a paired stimulus paradigm. The motor threshold (MT) was first established. The conditioning stimulus (70% MT) followed by the test stimulus (120% MT) was delivered at 100 ms for long ICI. Each run consisted of 10 trials, and the amplitude ratio of the mean conditioned Motor Evoked Potential (MEP) to control MEP was determined. A larger amplitude ratio indicates greater cortical excitability. The differences between Placebo and Baseline, and SGS and Baseline were obtained. These values were averaged across individuals to report a mean.
Time Frame: Baseline and Six months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio of MEP amplitude
Arm/Group | Placebo | Study Drug
Number analyzed (Participants) | 15 | 17
ratio of MEP amplitude | -9.3 (112.0) | 0.3 (98.6)

6. Secondary Outcome: Results of Physical Examination at the End of the Study Drug and Placebo Treatment Periods
Description: A physical examination was administered by a physician to subjects at the end of each six month treatment period, i.e., following completion of a six month period on SGS-742 or Placebo. Results of the examination ranged from 0-4 with scores defined as follows: 0=No observation; 1=Stable baseline findings; 2=New asymptomatic finding; 3=Patient reports some worsening of a baseline daily function associated with new finding; 4=Patient unable to carry out a baseline daily function associated with new finding
Time Frame: Six months
Population: One subject withdrew prior to end of Phase 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Study Drug
Number analyzed (Participants) | 18 | 18
Participants
  0 | 0 | 0
  1 | 14 | 15
  2 | 4 | 3
  3 | 0 | 0
  4 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a 16-21 month time period which included a 6 month +/- 2 week Phase 1 period, a 9 week +/- 2 week Washout period, a 6 month +/- 2 week Phase 2 period, followed by a 9 week +/- Washout period.
Groups:
- Placebo: Participants with SSADH Deficiency while on placebo for six months
  Placebo
- Washout Period Following Placebo: Participants with SSADH Deficiency having received Placebo, during the 9 week washout period
- Study Drug: Participants with SSADH Deficiency receiving SGS-742 while on study drug for six months
  SGS-742
- Washout Period Following Study Drug: Participants with SSADH Deficiency having received SGS-742, during the 9 week washout period
Arm/Group | Placebo | Washout Period Following Placebo | Study Drug | Washout Period Following Study Drug
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/16 | 0/19 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/16 | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 16/18 | 3/16 | 18/19 | 6/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=18) | Washout Period Following Placebo (N=16) | Study Drug (N=19) | Washout Period Following Study Drug (N=18)
Abdominal Pain (Gastrointestinal disorders) | 2 (3) | 0 (0) | 4 (6) | 1 (1)
Abnormal Urinary Analysis results (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Allergic Rhinitis (Ear and labyrinth disorders) | 1 (2) | 2 (2) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Anorexia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blister in the oral cavity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Concentration Impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 5 (5) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 2 (2) | 0 (0) | 3 (4) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Head lice (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperactivity (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Increased appetite (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Irritability (Psychiatric disorders) | 2 (5) | 0 (0) | 3 (3) | 2 (2)
Labile (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Labile (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 0 (0) | 2 (3) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Priapism (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 4 (4) | 1 (1)
Red eyes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizures (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sleepiness (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Strep throat (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (2) | 1 (1) | 2 (3) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1) | 2 (3) | 0 (0)
Weight gain (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/67/NCT02019667/Prot_SAP_000.pdf